CLINICAL TRIAL: NCT02756546
Title: Circulating MicroRNAs in Understanding Pathogenesis of Systemic Lupus Erythematosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Kortam, Teaching Assistant at faculty of Pharmacy Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BC (1016)
Record Dates: First submitted 2016-04-26; First posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Systemic Lupus Erythematosis
MeSH Terms: interventions — Cyclophosphamide; Hydroxychloroquine; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Healthy volunteers
- Patients (Active Comparator): SLE patients further divided into mild and severe patients
  Interventions: Drug: Cyclophosphamide; Drug: Hydroxychloroquine; Drug: Hydrocortisone

INTERVENTIONS:
Drug: Cyclophosphamide
  Arms: Patients
Drug: Hydroxychloroquine
  Arms: Patients
Drug: Hydrocortisone
  Arms: Patients

SUMMARY:
This study aims to identify the expression signature of miR-181a, miR-196a and miR-21 in plasma of SLE patients and difference in their expression among groups with different systemic lupus erythematosis disease activity index (SLEDAI) scores.

ELIGIBILITY:
Inclusion Criteria:

* Adult systemic lupus erythematosis patients

Exclusion Criteria:

* Patients younger than 18 years, patients with other autoimmune diseases or malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
MicroRNAs expression level | 3 months

IPD SHARING:
Plan to Share IPD: Yes
Publication